CLINICAL TRIAL: NCT06405841
Title: Costal Fracture Assessment for Relief and Enhancement of Quality of Life - CARE Study
Brief Title: Costal Fracture Assessment for Relief and Enhancement of Quality of Life
Acronym: CARE
Status: Not yet recruiting | Type: Observational
Sponsor: Ospedali Riuniti Trieste (Other)
Responsible Party: Principal Investigator, Manuela Mastronardi, Principal Investigator, Ospedali Riuniti Trieste
Other Study IDs: 345_2024H
Record Dates: First submitted 2024-05-04; First posted 2024-05-09 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Rib Fractures; Rib Trauma
MeSH Terms: conditions — Rib Fractures | interventions — Surveys and Questionnaires; Pain Management

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with rib fractures: Patients with rib fractures that correspond to inclusion and exclusion criteria
  Interventions: Other: Survey; Other: Pain management

INTERVENTIONS:
Other: Survey — All patients will be asked to complete a survey at 1, 2, 4, 12 and 24 weeks from the trauma to assess their quality of life
Other: Pain management — All patients will be asked about their pain management at 1, 2, 4, 12 and 24 weeks from the trauma to assess if they are under medication and what kind of medication are they taking

SUMMARY:
This study explores the impact of rib fractures on patient well-being and quality of life, aiming to identify effective interventions for pain relief and functional improvement. It investigates the long-term outcomes of conservative treatment for rib fractures, analyzing factors such as analgesic therapy, hospitalization duration, and respiratory infection rates. Anticipated results include a comprehensive assessment of patient quality of life and the potential translational implications for healthcare practice. Furthermore, the study aims to inform healthcare resource optimization, potentially guiding treatment decisions and improving patient outcomes within the National Health Service.

DETAILED DESCRIPTION:
Thoracic trauma remains a significant cause of morbidity and mortality in the traumatized population. Rib fractures are the most commonly encountered injuries after thoracic trauma, accounting for approximately 10-15% of all trauma-related hospital admissions. Fractured ribs serve as surrogate indicators of severe injuries, as most patients suffer additional critical injuries. Rib fractures are associated with significant long-term morbidity and disability, resulting in enduring physical impairment, dyspnea, and delayed return to normal daily and work activities, leading to decreased quality of life. Additionally, previous studies have demonstrated that up to a quarter of patients with rib fractures experience persistent chest pain even one year or more after the trauma. In current clinical practice, surgical treatment of rib fractures is increasingly common, as restoring chest wall integrity appears to alleviate pain and preserve normal breathing mechanics. While recent studies suggest that rib fracture fixation may improve lung function, reduce (pulmonary) complication rates, and shorten hospitalization and intensive care unit (ICU) stays in selected patients, a definitive consensus on which patients should undergo surgery has yet to be established. Contributing to the difficulty in determining optimal treatment for patients with rib fractures is the limited research on long-term quality of life and functional outcomes after rib fracture fixation or conservative management. Therefore, this study aims to investigate the quality of life of patients with rib fractures treated conservatively using a dedicated questionnaire and evaluate the type of analgesic medical therapy used, length of hospital stay, and rate of respiratory infections.

Expected Results, Translatability, and Impact on the National Health Service (SSN):

Expected Results: It is anticipated that the study will provide a detailed assessment of the quality of life of patients with rib fractures treated conservatively and their long-term quality of life. Additionally, the study aims to identify the most effective types of analgesic medical therapies in controlling rib fracture-related pain, as well as the duration of hospitalization and rate of respiratory infections associated with conservative treatment.

Translatability: The study results could have broad practical applications in the healthcare sector, providing guidance on best practices for rib fracture treatment. This could lead to greater efficacy in rib fracture management protocols, reducing or increasing the need for surgical interventions to improve patient quality of life.

Impact on the National Health Service (SSN): The study could have a significant impact on the SSN by providing evidence to optimize healthcare resources through more targeted management of rib fractures. If the results demonstrate that conservative treatment is ineffective for certain types of rib fractures, as it entails a longer hospital stay with very late return to daily and work activities, these patients could be selected for surgical treatment, resulting in savings for the SSN and an improvement in patient quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with rib fractures

Exclusion Criteria:

* cognitive impairment
* chronic pain due to pathologic fractures
* active cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients with rib fractures matching inclusion and exclusion criteria will be involved in the study
Sampling Method: Non-Probability Sample
Enrollment: 950 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Ability to achieve daily living activities (yes/no) | 1, 2, 4, 12 and 24 weeks from the trauma
  the ability to achieve daily living activities will be measured using a specific survey

SECONDARY OUTCOMES:
Pain killers assumption | 1, 2, 4, 12 and 24 weeks from the trauma
  evaluation of pain killers assumption (yes/no)
Respiratory infection rate | 1, 2, 4, 12 and 24 weeks from the trauma
  Incidence of respiratory infection in patients with rib fractures
Lenght of stay | to 2 years after the trauma
  Lenght of hospitalization in days

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - Emergency Department, Trieste, Italy
  - Intensive Care Unit, Trieste, Italy
  - Department of General Surgery, Trieste, TS
  - Department of Thoracic Surgery, Trieste, TS

REFERENCES:
- [Derived] Mastronardi M, Troian M, Germani P, Lovadina S, de Manzini N, Celaj E, Biloslavo A. Costal fracture assessment for relief and enhancement of quality of life-CARE study. Eur J Trauma Emerg Surg. 2025 Jan 9;51(1):3. doi: 10.1007/s00068-024-02689-3. PMID 39786597